CLINICAL TRIAL: NCT00447707
Title: Positive Choice: Prevention for Positive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R01DA015016 (NIH)
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-03

CONDITIONS: HIV Infections; Sexual Risk Behavior; Substance Use Risks
Keywords: Substance use; Unprotected sex; Behavioral intervention; HIV care; Prevention with Positives; HIV seronegativity
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Unsafe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Positive Choice

SUMMARY:
This is a randomized, controlled trial of Positive Choice, an interactive multimedia computer program, to determine whether it can detect and reduce risky behaviors among HIV-positive adults. The behaviors of interest are: unprotected anal or vaginal intercourse, illicit drug use, risky alcohol drinking, and failure to disclose HIV status to sex partners. The Positive Choice program is integrated into the routine operations of outpatient HIV clinics, where participating patients complete an in-depth risk assessment (computerized health questionnaire) before a regularly scheduled medical appointment. Participants assigned to the intervention arm receive brief, interactive risk-reduction counseling by an actor-portrayed Video Doctor and an educational worksheet. Their health care provider receives as summary cueing sheet, alerting them to the patient's risky behavior and readiness to change. Control participants complete the computerized risk assessment and receive the clinic's usual care. Three months after a baseline visit, intervention and control group patients are invited back to complete an additional risk assessment. The intervention group also receives a "booster" intervention. Six months after baseline, both groups complete a final risk assessment.

DETAILED DESCRIPTION:
A preliminary analysis of baseline data was conducted in January 2006, which indicated that the Positive Choice intervention achieved significant reductions in drug use. These findings were reported in a poster presentation at the XVI International AIDS Conference in Toronto, Canada, in August 2006. A final analysis of outcomes data was conducted in fall 2006 (September - December). Aggregate results from all five study sites are summarized below.

We found a high prevalence of risky behaviors in our sample (497/918, or 54%) and achieved high retention for follow-up in both groups (>80%). We found significant elimination of any drug use in the intervention group at both follow-ups. Among all participants who reported drug use at baseline, 66% of intervention participants continued their drug use at 3-month follow-up compared to 85% of control participants (OR 0.356, p<0.01). At 6-month follow-up, 59% of intervention participants continued their drug use compared to 88% of the control group (<0.001). Among participants who reported methamphetamine use at baseline, 58% continued their methamphetamine use at 3-month follow-up compared to 83% of control participants (OR 0.285, p=0.02). At 6-month follow-up, 53% of intervention participants continued their methamphetamine use compared to 73% of the control group (OR 0.344, p=0.03). We also found significantly less unprotected sex with casual partners by intervention participants at 3-month follow up (69% vs. 87%, OR 0.313, p=0.04), and fewer intervention participants who exceeded the recommended number of drinks per week at 3-months (53% vs. 78%, OR 0.310, p=0.02) Our findings indicate that the Positive Choice program was effective at reducing important behavioral risks among HIV-positive adults in care. Positive Choice is an appropriate and effective adjunct to routine medical care for HIV-positive adults.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* HIV-positive 3 months or longer,
* English speaking; and
* Receiving medical care at a participating clinic.

Exclusion Criteria:

* Less than 18 years old,
* HIV-positive less than 3 months,
* Non-English speaking; and
* Not receiving medical care at a participating clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 497
Dates: Start 2003-12; Study Completion 2006-09

PRIMARY OUTCOMES:
Elimination of risky drinking, illicit alcohol use, unprotected sex, and non-disclosure of HIV status to sex partners.

SECONDARY OUTCOMES:
Measures of change in risky alcohol use, illicit drug use, unprotected sex, and non-disclosure of HIV status to sex partners.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gerbert, PhD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - Adult Immunology Clinic, Highland Hospital, Oakland, California
  - AIDS Project East Bay (APEB), Oakland, California
  - East Bay AIDS Center (EBAC), Alta Bates Hospital, Oakland, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Adult Immunology Clinic, Fairmont Hospital, San Leandro, California

REFERENCES:
- [Background] Gerbert B, Danley DW, Herzig K, Clanon K, Ciccarone D, Gilbert P, Allerton M. Reframing "prevention with positives": incorporating counseling techniques that improve the health of HIV-positive patients. AIDS Patient Care STDS. 2006 Jan;20(1):19-29. doi: 10.1089/apc.2006.20.19. PMID 16426152
- [Derived] Gilbert P, Ciccarone D, Gansky SA, Bangsberg DR, Clanon K, McPhee SJ, Calderon SH, Bogetz A, Gerbert B. Interactive "Video Doctor" counseling reduces drug and sexual risk behaviors among HIV-positive patients in diverse outpatient settings. PLoS One. 2008 Apr 23;3(4):e1988. doi: 10.1371/journal.pone.0001988. PMID 18431475